CLINICAL TRIAL: NCT03057470
Title: Optimal Insulin Correction Factor in Post- High Intensity Exercise Hyperglycemia in Adults With Type 1 Diabetes: The FIT Study
Brief Title: Optimal Insulin Correction Factor in Post- High Intensity Exercise Hyperglycemia in Adults With Type 1 Diabetes (FIT)
Acronym: FIT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FIT
Record Dates: First submitted 2016-12-23; First posted 2017-02-20 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes; Exercise; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Motor Activity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0% Bolus Insulin Correction (Active Comparator): 0% Bolus Insulin Correction
  Interventions: Other: 0% bolus insulin correction
- 50% Bolus Insulin Correction (Active Comparator): 50% Bolus Insulin Correction
  Interventions: Drug: 50% bolus insulin correction
- 100% Bolus Insulin Correction (Active Comparator): 100% Bolus Insulin Correction
  Interventions: Drug: 100% bolus insulin correction
- 150% Bolus Insulin Correction (Active Comparator): 150% Bolus Insulin Correction
  Interventions: Drug: 150% bolus insulin correction

INTERVENTIONS:
Drug: 50% bolus insulin correction — Patients will receive 50% of their usual bolus insulin correction for post-exercise hyperglycemia
  Arms: 50% Bolus Insulin Correction
Drug: 100% bolus insulin correction — Patients will receive 100% of their usual bolus insulin correction for post-exercise hyperglycemia
  Arms: 100% Bolus Insulin Correction
Drug: 150% bolus insulin correction — Patients will receive 150% of their usual bolus insulin correction for post-exercise hyperglycemia
  Arms: 150% Bolus Insulin Correction
Other: 0% bolus insulin correction — Patients will receive no bolus insulin correction for post-exercise hyperglycemia
  Arms: 0% Bolus Insulin Correction

SUMMARY:
The overall objective of this study is to investigate the glycemic response of a 0%, 50%, 100% and 150% bolus insulin correction (based on personal insulin correction factor) of post-exercise hyperglycemia in physically active adults with type 1 diabetes (T1D) using multiple daily injections (MDI) in a controlled, but clinically representative, experimental setting.

DETAILED DESCRIPTION:
FIT is an open-label, repeated measures cross-over study. The overall objective of this study is to investigate the glycemic response of a 0%, 50%, 100% and 150% bolus insulin correction (based on personal insulin correction factor) of post-exercise hyperglycemia in physically active adults with type 1 diabetes (T1D) using multiple daily injections (MDI) in a controlled, but clinically representative, experimental setting. Following a 2 week screening phase, patients will enter an 8 week transition to insulin glargine U300 (Toujeo®) if on another basal insulin, in order to optimize their insulin dose and determine their individual insulin correction factor. The final phase of the study is the intervention phase, which consists of 4 separate visits. At each visit, the patient will perform 15 minutes of high intensity exercise in the morning. If they become hyperglycemic following exercise (blood glucose >8.0 mmol/L), they will receive one of four insulin correction doses (0% 50%, 100%, or 150% of their usual correction factor) in a randomized order. They will be monitored in the clinical pharmacology unit by study staff for the rest of the day and overnight. The patient will wear a continuous glucose monitor (CGM) during each intervention visit. The primary outcome of the study is the greatest net reduction in plasma glucose (YSI) following a 50%, 100% and 150% bolus insulin correction of post-exercise hyperglycemia, compared to no bolus insulin correction. Key secondary outcomes include the mean time spent in post-exercise hyperglycemia (>8.0 mmol/L), post-exercise euglycemia (4.0-8.0 mmol/L) and post-exercise hypoglycaemia (≤ 3.9 mmol/L) within 180 minutes and 24 hours following bolus insulin correction.

ELIGIBILITY:
Inclusion Criteria

* Male or female
* Clinical diagnosis of presumed autoimmune T1D
* Age 18-55 years, inclusive
* Duration of T1D ≥ 6 months
* Using MDI therapy for at least 6 months
* Fasting C-peptide value of < 0.7 ng/mL (0.23 nmol/L) at screening visit
* Patient must be willing to undergo an 8-week run-in phase prior to the study period where they will be required to use MDI therapy at least 4 times per day, and switch from their usual basal insulin to insulin glargine U300
* Exercise regularly: i.e. ≥ 30 minutes of moderate or vigorous aerobic activity ≥ 3 times/week for a minimum of 90 minutes weekly
* VO2peak ≥32 ml/kg/min for females and ≥ 35 ml/kg/min for males
* HbA1c between 6.0-9.0% inclusive at screening visit.
* Insulin total daily dose (TDD) ≥ 30 U/day
* In good general health with no known conditions that could influence the outcome of the trial, and in the judgement of the Investigator is a good candidate for the study based on review of available medical history, physical examination and clinical laboratory evaluations
* Willing to adhere to the protocol requirements for the duration of the study

Exclusion Criteria

* Pregnant or lactating
* Active diabetic retinopathy (proliferative diabetic retinopathy, or vitreous haemorrhage in past 6 months) that could potentially be worsened by the exercise protocol
* Any evidence of unstable cardiovascular disease, disorders or abnormalities as per physician's discretion. .
* Currently following a very low calorie or other weight-loss diet which may impact glucose control and mask the primary and secondary outcome measures
* More than one episode of severe hypoglycemia with seizure, coma or requiring assistance of another person during the past 6 months
* Known hypoglycemia unawareness
* Use of acetaminophen (Tylenol) during the run-in phase or study period
* Medications other than insulin that might impact outcome measures:
* Beta blockers
* Agents that affect hepatic glucose production such as beta adrenergic agonists and antagonists, xanthine derivatives
* Pramlintide
* Any non-insulin diabetes therapy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Reduction In Plasma Glucose (YSI) | 147 days

SECONDARY OUTCOMES:
Investigate Glycemic Response of a 0%, 50%, 100% and 150% Bolus Insulin Correction of Post-exercise Hyperglycemia Compared to no Bolus Insulin Correction | 147 days

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Aronson, MD, Principal Investigator — LMC Diabetes & Endocrinology
Locations (1):
- LMC Bayview, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Only overall study data will be shared

REFERENCES:
- [Background] 1. Robertson K, Adolfsson P, Scheiner G, Hanas R, Riddell M. Exercise in children and adolescents with diabetes. Pediatric diabetes. 2009;10(Journal Article):154. 2. Wasserman DH, Zinman B. Exercise in individuals with IDDM. Diabetes Care. 1994;17(8):924-937. 3. Galassetti P, Riddell MC. Exercise and type 1 diabetes (T1DM). Compr Physiol. 2013;3(3):1309-1336. 4. Zaharieva DP, Riddell MC. Prevention of exercise-associated dysglycemia: a case study-based approach. Diabetes Spectr. 2015;28(1):55-62. 5. Pivovarov JA, Taplin CE, Riddell MC. Current perspectives on physical activity and exercise for youth with diabetes. Pediatr Diabetes. 2015. 6. Marliss EB, Vranic M. Intense exercise has unique effects on both insulin release and its roles in glucoregulation: implications for diabetes. Diabetes. 2002;51 Suppl 1:S271-283. 7. Fahey AJ, Paramalingam N, Davey RJ, Davis EA, Jones TW, Fournier PA. The effect of a short sprint on postexercise whole-body glucose production and utilization rates in individuals with type 1 diabetes mellitus. J Clin Endocrinol Metab. 2012;97(11):4193-4200. 8. Benbenek-Klupa T, Matejko B, Klupa T. Metabolic control in type 1 diabetes patients practicing combat sports: at least two-year follow-up study. Springerplus. 2015;4:133. 9. Iscoe KE, Riddell MC. Continuous moderate-intensity exercise with or without intermittent high-intensity work: effects on acute and late glycaemia in athletes with Type 1 diabetes mellitus. Diabetic Med. 2011;28(7):824-832. 10. Graveling AJ, Frier BM. Risks of marathon running and hypoglycaemia in Type 1 diabetes. Diabet Med. 2010;27(5):585-588. 11. Tanenberg RJ, Newton CA, Drake AJ. Confirmation of hypoglycemia in the
- [Derived] Potashner D, Brown RE, Li A, Riddell MC, Aronson R. Paradoxical Rise in Hypoglycemia Symptoms With Development of Hyperglycemia During High-Intensity Interval Training in Type 1 Diabetes. Diabetes Care. 2019 Oct;42(10):2011-2014. doi: 10.2337/dc19-0609. Epub 2019 Aug 7. PMID 31391201
- [Derived] Aronson R, Brown RE, Li A, Riddell MC. Optimal Insulin Correction Factor in Post-High-Intensity Exercise Hyperglycemia in Adults With Type 1 Diabetes: The FIT Study. Diabetes Care. 2019 Jan;42(1):10-16. doi: 10.2337/dc18-1475. Epub 2018 Nov 19. PMID 30455336